CLINICAL TRIAL: NCT04576455
Title: A Phase II, Randomized, Open-Label, Multicenter Study Evaluating the Efficacy and Safety of GDC-9545 Compared With Physician's Choice of Endocrine Monotherapy in Patients With Previously Treated Estrogen Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study Evaluating the Efficacy and Safety of Giredestrant Compared With Physician's Choice of Endocrine Monotherapy in Participants With Previously Treated Estrogen Receptor-Positive, HER2-Negative Locally Advanced or Metastatic Breast Cancer (acelERA Breast Cancer)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO42312; 2020-001984-10 (EudraCT Number)
Record Dates: First submitted 2020-09-30; First posted 2020-10-06 (Actual); Results first posted 2023-03-10 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-12

CONDITIONS: Estrogen Receptor-Positive, HER2-Negative, Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — giredestrant; Fulvestrant; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Giredestrant (Experimental)
  Interventions: Drug: Giredestrant; Drug: LHRH Agonist
- Physician Choice of Endocrine Monotherapy (Active Comparator): The physician choice of endocrine monotherapy will be limited to fulvestrant or an aromatase inhibitor.
  Interventions: Drug: Fulvestrant or an Aromatase Inhibitor (Physician Choice); Drug: LHRH Agonist

INTERVENTIONS:
Drug: Giredestrant — Giredestrant is taken orally once per day on Days 1-28 of each 28-day cycle.
  Other Names: GDC-9545; RO7197597; RG6171
  Arms: Giredestrant
Drug: Fulvestrant or an Aromatase Inhibitor (Physician Choice) — Physician choice of endocrine monotherapy (fulvestrant or an aromatase inhibitor) is taken in accordance with the local prescribing information for the respective product.
  Arms: Physician Choice of Endocrine Monotherapy
Drug: LHRH Agonist — Only premenopausal/perimenopausal participants and male participants will receive a luteinizing hormone-releasing hormone (LHRH) agonist on Day 1 of each 28-day treatment cycle. The investigator will determine and supply the appropriate LHRH agonist locally approved for use in breast cancer.

SUMMARY:
This Phase II, randomized, open-label, multicenter study will evaluate the efficacy and safety of giredestrant compared with physician's choice of endocrine monotherapy in participants with estrogen receptor (ER)-positive, human epidermal growth factor receptor 2 (HER2)-negative locally advanced or metastatic breast cancer who have received one or two prior lines of systemic therapy in the locally advanced or metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Women who are postmenopausal or premenopausal/perimenopausal
* For women who are premenopausal or perimenopausal and for men: willing to undergo and maintain treatment with approved LHRH agonist therapy for the duration of study treatment
* Locally advanced or metastatic adenocarcinoma of the breast, not amenable to treatment with curative intent
* Documented ER-positive tumor and HER2-negative tumor, assessed locally
* Disease progression after treatment with one or two lines of systemic therapy (but not more than one prior targeted therapy) in the locally advanced or metastatic setting
* Measurable disease as defined per RECIST v.1.1 or bone only disease which must have at least one predominantly lytic bone lesion confirmed by CT or MRI which can be followed
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Adequate organ function

Exclusion Criteria:

* Prior treatment with a selective estrogen receptor degrader (SERD), with the exception of fulvestrant, if fulvestrant treatment was terminated at least 28 days prior to randomization
* Treatment with any investigational therapy within 28 days prior to randomization
* Advanced, symptomatic, visceral spread that is at risk of life-threatening complications
* Known active uncontrolled or symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease
* Active cardiac disease or history of cardiac dysfunction
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2020-11-27 (Actual); Primary Completion 2022-02-18 (Actual); Study Completion 2027-08-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (85):
- United States (3):
  - Northwest Georgia Oncology Centers PC - Marietta, Marietta, Georgia
  - University Hospitals Seidman Cancer Center, Cleveland, Ohio
  - Northwest Cancer Specialists - Portland (SW Barnes Rd), Tigard, Oregon
- Argentina (5):
  - Instituto Angel Roffo, Buenos Aires
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Fundación Scherbovsky, Mendoza
  - Hosp Provincial D. Centenarios, Rosario
  - Organizacion Medica de Investigacion, San Nicolás
- Australia (2):
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Sunshine Hospital, St Albans, Victoria
- Brazil (5):
  - Pronutrir - suporte nutricional e quimioterapia ltda., Fortaleza, Ceará
  - Oncosite - Centro de Pesquisa Clinica Em Oncologia Ltda, Ijuí, Rio Grande do Sul
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo, São Paulo
- China (10):
  - The First Hospital of Jilin University, Changchun
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Linyishi Cancer Hospital, Linyi
  - The Third Hospital of Nanchang, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an
  - Zhejiang Cancer Hospital, Zhejiang
- Germany (5):
  - Hämato-Onkologische Schwerpunktpraxis am Klinikum Aschaffenburg, Aschaffenburg
  - Frauenarzt-Zentrum Zehlendorf an der Teltower Eiche, Berlin
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - St. Vincenz-Krankenhaus Paderborn, Paderborn
  - Gynäkologie Kompetenzzentrum, Stralsund
- Israel (3):
  - Assuta Medical Center- Ashdod, Ashdod
  - Hadassah Ein Karem Hospital, Jerusalem
  - Meir Medical Center, Kfar Saba
- Poland (3):
  - Bialostockie Centrum Onkologii, Bialystok
  - Narodowy Instytut Onkologii Odzia? w Gliwicach, Gliwice
  - Narodowy Inst.Onkologii im.Sklodowskiej-Curie Panstw.Inst.Bad, Warsaw
- Russia (10):
  - Krasnoyarsk Regional Oncology Dispensary n.a. Krizhanovsky, Krasnoyarsk, Krasnodarskiy Kray
  - Petrov Research Inst. of Oncology, Pesochny, Leningrad
  - Blokhin Cancer Research Center, Moskva, Moscow Oblast
  - Filial #1 Regional Oncology Dispensary of Nizhniy Novgorod, Nizhny Novgorod, Niznij Novgorod
  - St. Petersburg SHI "City Clinical Oncology Dispensary", Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary of Ministry of Healthcare of Tatarstan Republic, Kazan', Tatarstan Republic
  - Clinical Oncology Centre # 1, Krasnodar
  - Multidisciplinary clinic Reaviz, Samara
  - Volgograd Regional Clinical Oncology Dispensary, Volgograd
  - Regional Clinical Oncology Hospital, Yaroslavl
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Africa (3):
  - Iatros International, Bloemfontein
  - Cancercare Langenhoven Drive Oncology Centre, Port Elizabeth
  - Eastleigh Breast Care Centre, Pretoria
- South Korea (8):
  - Soon Chun Hyang University Cheonan Hospital, Dongnam-gu, Cheonan-si
  - National Cancer Center, Goyang-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
- Taiwan (5):
  - Changhua Christian Hospital, Changhua
  - National Cheng Kung Uni Hospital, Tainan
  - Chi-Mei Medical Centre, Tainan
  - Veterans General Hospital, Taipei
  - Chang Gung Memorial Hosipital at Linkou, Taoyuan Hsien
- Thailand (5):
  - Chulalongkorn Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai Hosp, Chang Mai
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (8):
  - Memorial Ankara Hastanesi, Ankara
  - Ankara City Hospital, Ankara
  - Memorial Antalya Hospital, Antalya
  - Dicle University Faculty of Medicine, Diyarbakır
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi, Istanbul
  - Prof. Dr. Cemil Tascioglu City Hospital, Istanbul
  - Katip Celebi University Ataturk Training and Research Hospital, Izmir
  - Medikal Park Samsun, Samsun
- Ukraine (4):
  - Zhytomyr Regional Oncology Center, Zhytomyr, KIEV Governorate
  - Kyiv City Clinical Oncological Center, Kyiv
  - MI Kyiv Regional Council Kyiv Regional Oncological Dispensary, Kyiv
  - RCI Sumy Regional Clinical Oncological Dispensary, Sumy
- United Kingdom (4):
  - Princess Alexandra Hospital, Harlow
  - Guys & St Thomas Hospital, London
  - Nottingham City Hospital, Nottingham
  - Peterborough City Hospital, Peterborough

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Martin M, Lim E, Chavez-MacGregor M, Bardia A, Wu J, Zhang Q, Nowecki Z, Cruz FM, Safin R, Kim SB, Schem C, Montero AJ, Khan S, Bandyopadhyay R, Moore HM, Shivhare M, Patre M, Martinalbo J, Roncoroni L, Perez-Moreno PD, Sohn J; acelERA Breast Cancer Study Investigators. Giredestrant for Estrogen Receptor-Positive, HER2-Negative, Previously Treated Advanced Breast Cancer: Results From the Randomized, Phase II acelERA Breast Cancer Study. J Clin Oncol. 2024 Jun 20;42(18):2149-2160. doi: 10.1200/JCO.23.01500. Epub 2024 Mar 27. PMID 38537155
- [Derived] Malhi V, Nowicka M, Chen YC, Agarwal P, Waldvogel M, Lien YTK, Hafner M, Perez-Moreno P, Moore HM, Yu J. UGT1A4 Polymorphism is not Associated with a Clinically Relevant Change in Giredestrant Exposure. Cancer Chemother Pharmacol. 2024 Jul;94(1):117-122. doi: 10.1007/s00280-023-04634-4. Epub 2024 Feb 2. PMID 38305868

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled in this study at 85 investigational sites in the following countries: Argentina, Australia, Brazil, China, Germany, Israel, Poland, Republic of Korea, Russian Federation, Singapore, South Africa, Taiwan, Thailand, Turkey, Ukraine, United Kingdom, and the United States. The study is ongoing.
Pre-assignment Details: A total of 303 participants were enrolled in this study, one of whom was randomized to the giredestrant arm and received fulvestrant in error and was grouped in the physician's choice of endocrine monotherapy (PCET) arm for safety analysis.
Groups:
- Giredestrant: Participants received giredestrant, 30 milligrams (mg), orally (PO), once daily (QD), on Days 1-28 (and luteinizing hormone-releasing hormone [LHRH] agonist according to clinical practice for the selected agent on Day 1 for pre/perimenopausal participants and male participants only) of each 28-day cycle until disease progression or unacceptable toxicity, whichever occurs first.
- Physician's Choice of Endocrine Monotherapy: Participants received physician's choice of endocrine monotherapy (PCET; fulvestrant or aromatase inhibitor) in accordance with the local prescribing information for the respective product (and LHRH agonist according to clinical practice for the selected agent on Day 1 of each 28-day cycle for premenopausal/perimenopausal participants and male participants only) until disease progression or unacceptable toxicity, whichever occurs first.
Period: Overall Study
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Started | 151 | 152
Safety-Evaluable Population (Safety-Evaluable Population included all participants who received at least one dose of the study treatment (giredestrant or PCET).) | 150 (1 participant randomized to the giredestrant arm received fulvestrant in error, and thus was counted in the PCET arm for safety analysis.) | 152 (1 participant randomized to the giredestrant arm received fulvestrant in error, and thus was counted in this arm for safety analysis. 1 participant randomized to this arm discontinued the study before receiving any study drug.)
Completed | 0 | 0
Not Completed | 151 | 152
Not completed — Ongoing in the Study | 48 | 58
Not completed — Death | 83 | 77
Not completed — Lost to Follow-up | 4 | 5
Not completed — Withdrawal by Subject | 16 | 12

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) included all participants assigned to treatment groups as randomized by the interactive voice or web-based response system (IxRS).
Groups:
- Giredestrant: Participants received giredestrant, 30 mg, PO, QD, on Days 1-28 (and LHRH agonist according to clinical practice for the selected agent on Day 1 for pre/perimenopausal participants and male participants only) of each 28-day cycle until disease progression or unacceptable toxicity, whichever occurs first.
- Total: Total of all reporting groups
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy | Total
Number analyzed (Participants) | 151 | 152 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (12.4) | 57.8 (10.7) | 58.6 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 151 | 151 | 302
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 23 | 20 | 43
  Not Hispanic or Latino | 128 | 132 | 260
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 58 | 66 | 124
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 89 | 81 | 170
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 2 | 3
Site of Disease (Visceral or Non-Visceral) [Count of Participants; unit: Participants] — Visceral disease was defined as any lung and/or liver involvement. Non-visceral disease was defined as the absence of any lung and/or liver involvement.
  Participants
    Visceral Disease | 109 | 110 | 219
    Non-visceral Disease | 42 | 42 | 84
Prior Treatment With CDK4/6 Inhibitor (Yes or No) [Count of Participants; unit: Participants]
  Yes, Prior Treatment With CDK4/6 Inhibitor | 63 | 62 | 125
  No Prior Treatment With CDK4/6 Inhibitor | 88 | 90 | 178
Prior Treatment With Fulvestrant (Yes or No) [Count of Participants; unit: Participants]
  Yes, Prior Treatment With Fulvestrant | 29 | 29 | 58
  No Prior Treatment With Fulvestrant | 122 | 123 | 245
Estrogen Receptor (ESR1) Mutation Status [Count of Participants; unit: Participants] — Baseline detectable ESR1 mutations present in circulating tumor DNA (ctDNA) were determined with next-generation sequencing from a pre-treatment plasma collection using the FoundationOne Liquid CDx assay conducted at Foundation Medicine.
  Participants
    ESR1 mutation detected | 51 | 39 | 90
    ESR1 no mutation detected | 66 | 76 | 142
    Not Evaluable | 34 | 37 | 71

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS), as Determined by the Investigator According to Response Evaluation Criteria in Solid Tumors, Version 1.1 (RECIST v1.1)
Description: PFS was defined as the Kaplan-Meier estimate of time from randomization to the first occurrence of disease progression as determined by the investigator according to RECIST v1.1, or death from any cause (whichever occurs first). Disease progression was defined as ≥20% increase in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions. Kaplan-Meier methodology was used to estimate median PFS. The 95% confidence interval for the median was computed using the method of Brookmeyer and Crowley. Participants without the occurrence of disease progression or death as of the clinical cutoff were censored at the time of the last tumor assessment prior to the clinical cutoff or at the time of randomization plus 1 day for those without post-baseline assessment.
Time Frame: From randomization to the first occurrence of disease progression or death from any cause, whichever occurs first (duration of follow-up, median [range]: 7.9 [0.0-14.1] months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
months | 5.55 [4.93 to 7.36] | 5.36 [3.71 to 5.55]
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Superiority; p = 0.1757, Log Rank; Stratified analysis (strata are: site of disease, prior CDK4/6i treatment, and prior fulvestrant treatment); Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.60 to 1.10] — Giredestrant vs. PCET

2. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the Kaplan-Meier estimate of time from randomization to death from any cause. Kaplan-Meier methodology was used to estimate median OS. The 95% confidence interval for the median was computed using the method of Brookmeyer and Crowley. Analysis strata are: Site of disease, Prior treatment with CDK4/6 inhibitor and Prior treatment with fulvestrant. Hazard ratios were estimated by Cox regression. Data for participants who were alive at the time of the analysis data cutoff were censored at the last date they were known to be alive. Data from participants without postbaseline information were censored at the date of randomization plus 1 day.
Time Frame: From randomization to death from any cause (duration of follow-up, median [range]: 34.6 [0.0-41.8] months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
Months | 27.50 [23.20 to 32.69] | 29.77 [26.78 to NA] — The upper limit of the 95% confidence interval (CI) was not evaluable because of an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Superiority; p = 0.3446, Log Rank; Stratified analysis (strata are: site of disease, prior CDK4/6i treatment, and prior fulvestrant treatment); Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.85 to 1.60] — Giredestrant vs. PCET

3. Secondary Outcome: Objective Response Rate, as Determined by the Investigator According to RECIST v1.1
Description: The objective response rate is defined as the percentage of participants with a complete response (CR) or partial response (PR) on two consecutive occasions at least 4 weeks apart. Per RECIST v1.1, CR is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must have reduction in short axis to <10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: From randomization until disease progression or death (up to approximately 15 months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
Percentage of participants | 12.6 [7.75 to 18.95] | 7.2 [3.67 to 12.58]
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Superiority; p = 0.1126, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.86 to 4.07] — Giredestrant vs. PCET
Statistical Analysis 2: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Superiority; Difference in Objective Response Rates = 5.35, 95% CI 2-sided [-1.97 to 12.78] — Giredestrant vs. PCET

4. Secondary Outcome: Duration of Response (DOR), as Determined by the Investigator According to RECIST v1.1
Description: DOR is defined as the Kaplan-Meier estimate of time from the first occurrence of a documented objective response to disease progression as determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first). Objective response rate is defined as the percentage of participants with a CR or PR on two consecutive occasions at least 4 weeks apart. Per RECIST v1.1, CR is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must have reduction in short axis to <10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR. Disease progression is defined as ≥20% increase in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions.
Time Frame: From first occurrence of documented objective response to disease progression or death from any cause, whichever occurs first (up to approximately 15 months)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 19 | 11
Months | NA [5.55 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event. | 7.39 [7.39 to NA] — The upper limit of the 95% CI was not evaluable because of an insufficient number of participants with the event.

5. Secondary Outcome: Clinical Benefit Rate, as Determined by the Investigator According to RECIST v1.1
Description: The clinical benefit rate is defined as the percentage of participants with stable disease for ≥24 weeks or a CR or PR. Per RECIST v1.1, CR is defined as disappearance of all target and non-target lesions. Any pathological lymph nodes must have reduction in short axis to <10 millimeters (mm). PR is defined as at least a 30% decrease in the sum of diameters of all target lesions, taking as reference the baseline sum of diameters, in the absence of CR.
Time Frame: From randomization until disease progression or death (up to approximately 15 months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
Percentage of participants | 31.8 [24.46 to 39.85] | 21.1 [14.87 to 28.40]
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Superiority; p = 0.0289, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.79, 95% CI 2-sided [1.06 to 3.04] — Giredestrant vs. PCET
Statistical Analysis 2: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Superiority; Difference in Clinical Benefit Rates = 10.74, 95% CI 2-sided [0.33 to 20.86] — Giredestrant vs. PCET

6. Secondary Outcome: Investigator-Assessed PFS, in Subgroups Categorized by Estrogen Receptor (ESR1) Mutation Status
Description: PFS was defined as the Kaplan-Meier estimate of time from randomization to the first occurrence of disease progression determined by the investigator according to RECIST v1.1 or death from any cause (whichever occurs first). Disease progression was defined as ≥20% increase in in the sum of diameters of target lesions, unequivocal progression in non-target lesions, and/or appearance of new lesions. Investigator-assessed PFS was analyzed in subgroups categorized by baseline ESR1 mutation status (i.e., with or without ESR1 mutation at baseline) from plasma circulating tumor deoxyribonucleic acid (ctDNA). Participants without the occurrence of disease progression or death as of the clinical cutoff were censored at the time of the last tumor assessment prior to the clinical cutoff or at the time of randomization plus 1 day for those without post-baseline assessment.
Time Frame: as for outcome 1
Population: ctDNA-evaluable population included all FAS participants with evaluable plasma ctDNA at baseline. Number analyzed is the number of participants with data available for analysis at the specified time point. Participants without the occurrence of disease progression or death as of the clinical cutoff were censored at the time of last tumor assessment prior to the clinical cutoff or at the time of randomization plus 1 day for those without post-baseline assessment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Physician's Choice of Endocrine Monotherapy: Participants received physician's choice of endocrine monotherapy (PCET; fulvestrant or aromatase inhibitor) in accordance with the local prescribing information for the respective product. In addition, premenopausal/perimenopausal participants and male participants received a LHRH agonist according to clinical practice for the selected agent on Day 1 of each 28-day treatment cycle until disease progression or unacceptable toxicity, whichever occurs first.
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 117 | 115
months
  PFS by ESR1 Mutation Detected at Baseline: number analyzed (Participants) | 51 | 39
  PFS by ESR1 Mutation Detected at Baseline | 5.32 [3.61 to 5.59] | 3.48 [1.81 to 3.81]
  PFS by ESR1 Mutation Not Detected at Baseline: number analyzed (Participants) | 66 | 76
  PFS by ESR1 Mutation Not Detected at Baseline | 7.20 [5.36 to 11.17] | 6.60 [5.32 to NA] — The upper limit of the 95% CI was not evaluable because of an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; This statistical analysis is done for PFS by ESR1 mutation detected at baseline; Test type: Superiority; p = 0.0610, Log Rank; Stratified analysis (strata are: site of disease, prior CDK4/6i treatment, and prior fulvestrant treatment); Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.35 to 1.03] — Giredestrant vs. PCET
Statistical Analysis 2: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; This statistical analysis is done for PFS by ESR1 Mutation not detected at baseline; Test type: Superiority; p = 0.5947, Log Rank; Stratified analysis (strata are: site of disease, prior CDK4/6i treatment, and prior fulvestrant treatment); Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.54 to 1.42] — Giredestrant vs. PCET

7. Secondary Outcome: Time to Deterioration (TTD) in Pain Severity, Based on the Brief Pain Inventory-Short Form (BPI-SF) Questionnaire
Description: TTD in pain severity is defined as time to first documented ≥2-point increase from Baseline in the "Worst Pain" item from the BPI-SF Questionnaire held for at least two consecutive cycles or an initial ≥2-point worsening followed by death or treatment discontinuation within 3 weeks from the last assessment. The BPI-SF is a self administered questionnaire developed to assess the severity of pain (the sensory dimension) as well as the degree to which pain interferes with function (the reactive dimension). The BPI-SF uses 10-point numeric rating scale, with 0="No pain", "No interference" to 10="Pain as bad as you can imagine", "Highest imaginable interference". A lower score indicates improvement. 95% CI for median was computed using the method of Brookmeyer and Crowley. Strata are: Site of disease, Prior treatment with CDK4/6 inhibitor, and Prior treatment with fulvestrant. Hazard ratios were estimated by Cox regression.
Time Frame: From Baseline until treatment discontinuation (up to approximately 41 months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
months | 28.65 [18.43 to NA] — The upper limit of the 95% CI was not evaluable because of an insufficient number of participants with the event. | NA [16.59 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Other; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.58 to 1.40] — Giredestrant vs. PCET

8. Secondary Outcome: TTD in Pain Presence and Interference, Based on the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ)-C30 Pain Scale Score
Description: TTD in pain presence and interference is defined as the time to first documented ≥10-point decrease from baseline in the EORTC QLQ-C30 linearly transformed pain scale score (0-100 scale) held for at least 2 consecutive cycles or an initial ≥10-point worsening followed by death or treatment discontinuation within 3 weeks from the last assessment. EORTC QLQ-C30 is a patient-reported measure with 30 questions assessing 5 aspects of functioning, 3 symptom scales, global health and quality of life, and 6 single items with a recall period of the previous week. The pain scale is scored on a 4-point scale (1=Not at All to 4=Very Much); higher scores indicate worse pain symptoms. The 95% CI for median was computed using the method of Brookmeyer and Crowley. Strata are: Site of disease, Prior treatment with CDK4/6 inhibitor, and Prior treatment with fulvestrant. Hazard ratios were estimated by Cox regression.
Time Frame: From Baseline until treatment discontinuation (up to approximately 41 months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
months | 22.14 [18.43 to NA] — The upper limit of the 95% CI was not evaluable because of an insufficient number of participants with the event. | NA [20.27 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.49 to 1.12] — Giredestrant vs. PCET

9. Secondary Outcome: TTD in Physical Functioning (PF), Based on the EORTC QLQ-C30 PF Scale Score
Description: TTD in PF is defined as the time to first documented ≥10-point decrease from baseline in the EORTC QLQ-C30 linearly transformed PF scale score (0-100 scale) held for at least 2 consecutive cycles or an initial ≥10-point worsening followed by death or treatment discontinuation within 3 weeks from the last assessment. EORTC QLQ-C30 is a patient-reported measure with 30 questions assessing 5 aspects of functioning, 3 symptom scales, global health and quality of life, and 6 single items with a recall period of the previous week. The PF scale has 5 questions scored on a 4-point scale (1=Not at All to 4=Very Much); higher scores indicate better function. The 95% CI for median was computed using the method of Brookmeyer and Crowley. Strata are: Site of disease, Prior treatment with CDK4/6 inhibitor, and Prior treatment with fulvestrant. Hazard ratios were estimated by Cox regression.
Time Frame: From Baseline until treatment discontinuation (up to approximately 41 months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
months | NA [28.65 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event. | NA [23.29 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Other; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.53 to 1.35] — Giredestrant vs. PCET

10. Secondary Outcome: TTD in Role Functioning (RF), Based on the EORTC QLQ-C30 RF Scale Score
Description: TTD in RF is defined as the time to first documented ≥10-point decrease from baseline in the EORTC QLQ-C30 linearly transformed RF scale score (0-100 scale) held for at least 2 consecutive cycles or an initial ≥10-point worsening followed by death or treatment discontinuation within 3 weeks from the last assessment. EORTC QLQ-C30 is a patient-reported measure with 30 questions assessing 5 aspects of functioning, 3 symptom scales, global health and quality of life, and 6 single items with a recall period of the previous week. The RF is scored on a 4-point scale (1=Not at All to 4=Very Much); higher scores indicate better function. The 95% CI for median was computed using the method of Brookmeyer and Crowley. Strata are: Site of disease, Prior treatment with CDK4/6 inhibitor, and Prior treatment with fulvestrant. Hazard ratios were estimated by Cox regression.
Time Frame: From Baseline until treatment discontinuation (up to approximately 41 months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
months | NA [18.43 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event. | NA [22.31 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Other; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.72 to 1.69] — Giredestrant vs. PCET

11. Secondary Outcome: TTD in Global Health Status and Quality of Life (GHS/QoL), Based on the EORTC QLQ-C30 GHS/QoL Scale Score
Description: TTD in GHS/QoL is defined as the time to first documented ≥10-point decrease from baseline in the EORTC QLQ-C30 linearly transformed RF scale score (0-100 scale) held for at least 2 consecutive cycles or an initial ≥10-point worsening followed by death or treatment discontinuation within 3 weeks from the last assessment. EORTC QLQ-C30 is a patient-reported measure with 30 questions assessing 5 aspects of functioning, 3 symptom scales, global health and quality of life, and 6 single items with a recall period of the previous week. The GHS/QoL scale has 7 possible scores of responses (1=very poor to 7=excellent); higher scores indicate better QoL. The 95% CI for median was computed using the method of Brookmeyer and Crowley. Strata are: Site of disease, Prior treatment with CDK4/6 inhibitor, and Prior treatment with fulvestrant. Hazard ratios were estimated by Cox regression.
Time Frame: From Baseline until treatment discontinuation (up to approximately 41 months)
Population: FAS included all participants assigned to treatment groups as randomized by the IxRS.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
Number analyzed (Participants) | 151 | 152
months | NA [31.38 to NA] — The median and the upper limit of the 95% CI were not evaluable because of an insufficient number of participants with the event. | NA [NA to NA] — The median and the 95% CI were not evaluable because of an insufficient number of participants with the event.
Statistical Analysis 1: Comparison: Giredestrant vs Physician's Choice of Endocrine Monotherapy; Test type: Other; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.47 to 1.18] — Giredestrant vs. PCET

12. Secondary Outcome: Number of Participants With Adverse Events (AEs), Severity Determined According to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 (NCI CTCAE v5.0)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product; any new disease or exacerbation of an existing disease; recurrence of an intermittent medical condition; any deterioration in a laboratory value or other clinical test; AEs that are related to a protocol-mandated intervention, including those that occur prior to assignment of study treatment.
Time Frame: From first dose until 30 days after final dose of study drug (up to approximately 55 months)
Reporting Status: Not Posted

13. Secondary Outcome: Number of Participants With Vital Sign Abnormalities Over the Course of the Study
Description: Vital signs include respiratory rate, pulse rate, systolic and diastolic blood pressure while the patient is in a seated position, and temperature.
Time Frame: Assessed at Baseline and predose on Day 1 of every cycle (1 cycle is 28 days) until 30 days after the final dose of study drug (up to approximately 55 months)
Reporting Status: Not Posted

14. Secondary Outcome: Number of Participants With Clinical Laboratory Test Abnormalities for Hematology Parameters Over the Course of the Study
Description: Hematology parameters include white blood cell (WBC) count, red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, and differential count (neutrophils, eosinophils, basophils, monocytes, lymphocytes, other cells).
Time Frame: as for outcome 13
Reporting Status: Not Posted

15. Secondary Outcome: Number of Participants With Clinical Laboratory Test Abnormalities for Biochemistry Parameters Over the Course of the Study
Description: Biochemistry parameters include bicarbonate or total carbon dioxide, sodium, potassium, chloride, glucose, blood urea nitrogen (BUN) or urea, creatinine, total protein, albumin, phosphate, calcium, total and direct bilirubin, alkaline phosphatase level test (ALP), Alanine transaminase (ALT), aspartate aminotransferase (AST), urate, and lactate dehydrogenase (LDH).
Time Frame: as for outcome 13
Reporting Status: Not Posted

16. Secondary Outcome: Plasma Concentration of Giredestrant at Specified Timepoints
Time Frame: Cycle 1 Day 1 3-hours postdose, Cycle 2 Day 1 predose, Cycle 2 Day 1 3-hour postdose, Cycle 3 Day 1 predose
Population: Pharmacokinetics (PK)-Evaluable Population: All randomized patients in the giredestrant arm who had at least one evaluable post-dose giredestrant plasma concentration. The overall number of participants analyzed is the total number of unique participants who had an evaluable PK sample for at least one timepoint. The number analyzed at a given timepoint indicates those with an evaluable sample for the specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/mL)
Arm/Group | Giredestrant
Number analyzed (Participants) | 148
nanograms per millilitre (ng/mL)
  Cycle 1 Day 1 3-hours postdose: number analyzed (Participants) | 139
  Cycle 1 Day 1 3-hours postdose | 117 (107)
  Cycle 2 Day 1 predose: number analyzed (Participants) | 135
  Cycle 2 Day 1 predose | 171 (64.5)
  Cycle 2 Day 1 3-hour postdose: number analyzed (Participants) | 132
  Cycle 2 Day 1 3-hour postdose | 268 (57.6)
  Cycle 3 Day 1 predose: number analyzed (Participants) | 112
  Cycle 3 Day 1 predose | 151 (68.5)

ADVERSE EVENTS:
Time Frame: For adverse events (AEs): From first dose of study drug until 30 days after the final dose of study drug (duration of treatment exposure, median [range]: giredestrant: 5.5 [0.9-40.8] months and PCET: 4.6 [0.03-37.1] months). For all-cause mortality: From randomization to death from any cause (duration of follow-up for both arms, median [range]: 34.6 [0.0-41.8] months). Data collection is ongoing and AEs will be updated within 1 year of the end of trial.
Description: All-cause mortality is reported for FAS which included all participants assigned to treatment groups as randomized by the IxRS.
  Serious and other AEs are reported for Safety-Evaluable Set which included all participants who received at least one dose of the study treatment (giredestrant or PCET). As pre-specified in the protocol, participants were grouped according to treatment received (giredestrant or PCET) for collection of AEs.
Arm/Group | Giredestrant | Physician's Choice of Endocrine Monotherapy
All-Cause Mortality (participants affected / at risk) | 83/151 | 77/152
Serious Adverse Events (participants affected / at risk) | 20/150 | 15/152
Other Adverse Events (participants affected / at risk) | 108/150 | 87/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Giredestrant (N=150) | Physician's Choice of Endocrine Monotherapy (N=152)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular graft stenosis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0)
Partial seizures (Nervous system disorders) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Giredestrant (N=150) | Physician's Choice of Endocrine Monotherapy (N=152)
Anaemia (Blood and lymphatic system disorders) | 18 (19) | 14 (15)
Constipation (Gastrointestinal disorders) | 12 (12) | 12 (15)
Diarrhoea (Gastrointestinal disorders) | 15 (19) | 6 (15)
Nausea (Gastrointestinal disorders) | 17 (26) | 13 (15)
Vomiting (Gastrointestinal disorders) | 15 (19) | 4 (7)
Asthenia (General disorders) | 12 (13) | 5 (5)
Chest pain (General disorders) | 10 (10) | 1 (1)
Fatigue (General disorders) | 14 (18) | 9 (10)
Product dose omission in error (Injury, poisoning and procedural complications) | 18 (41) | 0 (0)
Alanine aminotransferase increased (Investigations) | 20 (29) | 13 (14)
Aspartate aminotransferase increased (Investigations) | 26 (34) | 17 (20)
Blood bilirubin increased (Investigations) | 10 (18) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 10 (12) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (23) | 18 (19)
Back pain (Musculoskeletal and connective tissue disorders) | 9 (11) | 6 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (11) | 10 (10)
Dizziness (Nervous system disorders) | 11 (12) | 8 (8)
Headache (Nervous system disorders) | 15 (20) | 15 (28)
Hypertension (Vascular disorders) | 10 (13) | 3 (4)
COVID-19 (Infections and infestations) | 8 (8) | 10 (10)
Product dose omission issue (Injury, poisoning and procedural complications) | 18 (44) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 8 (16) | 5 (5)
Blood creatinine increased (Investigations) | 8 (9) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8) | 10 (12)
Hot flush (Vascular disorders) | 9 (9) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04576455/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-27): https://cdn.clinicaltrials.gov/large-docs/55/NCT04576455/SAP_001.pdf